CLINICAL TRIAL: NCT00064805
Title: Cognitively-based Treatments of Acquired Dyslexias
Brief Title: Therapy for Reading Problems in Adults After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD036019 (NIH)
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-04

CONDITIONS: Dyslexia, Acquired; Brain Injuries; Cerebrovascular Accident
Keywords: Cognitive therapy; Aphasia therapy; Alexia; Acquired dyslexia; Phonological deficits; Orthographic deficits; Brain disorders; Brain injury; Stroke
MeSH Terms: conditions — Dyslexia, Acquired; Brain Injuries; Stroke; Dyslexia; Brain Diseases

INTERVENTIONS:
Behavioral: Cognitive Therapy to Improve Reading

SUMMARY:
Adults who sustain brain damage due to stroke, head injury, or traumatic surgery may develop difficulty reading. This study examines the effectiveness of behavior-based programs to improve reading ability in these individuals.

DETAILED DESCRIPTION:
Acquired disorders of reading (acquired dyslexia) are common in patients with aphasia subsequent to left hemisphere stroke. Even when language functions recover sufficiently to enable the patient to return to work, continuing dyslexia often interferes significantly with job performance. This study will evaluate cognitive therapies for the treatment of acquired dyslexia.

Each therapy is based upon a cognitive neuropsychological model of reading; the therapies target specific types of reading deficit and stem from the question of re-learning versus re-organization of function. The therapies focus on dyslexic disorders stemming from the following underlying deficits: 1) impaired access to the orthographic word form from the visual modality (pure alexia); 2) impaired orthographic/phonologic connections (phonologic/deep dyslexia); and 3) decreased ability to hold phonologic codes in memory (phonologic text alexia).

Participants in this study will undergo a comprehensive and detailed battery of reading and reading-related tests to determine the underlying impairment causing the reading deficit. Based upon the results of these tests, the patient's dyslexic disorder will be characterized and, if appropriate, the patient will be assigned to one of the treatment programs devised specifically for that type of deficit. Treatment programs are evaluated for efficacy by comparing the accuracy and speed of reading pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria

* Reading deficit subsequent to stroke, traumatic brain injury, brain surgery, or other brain damage
* Ability to attend 2-3 sessions per week for several months at Georgetown University in Washington, DC

Exclusion Criteria

* History of developmental dyslexia or learning disabilities
* Best corrected vision less than 20/40
* Less than 10 years of formal education
* Significant memory or comprehension problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Improved accuracy and/or speed of reading individual words aloud.

SECONDARY OUTCOMES:
Improved accuracy and/or speed of reading text aloud.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda B. Friedman, Ph.D., Principal Investigator — Georgetown University Medical School
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Friedman RB, Lott SN. Rapid word identification in pure alexia is lexical but not semantic. Brain Lang. 2000 May;72(3):219-37. doi: 10.1006/brln.2000.2286. PMID 10764518
- [Background] Nitzberg Lott S, Friedman RB. Can treatment for pure alexia improve letter-by-letter reading speed without sacrificing accuracy? Brain Lang. 1999 May;67(3):188-201. doi: 10.1006/brln.1999.2054. PMID 10210630
- [Background] Friedman RB, Sample DM, Lott SN. The role of level of representation in the use of paired associate learning for rehabilitation of alexia. Neuropsychologia. 2002;40(2):223-34. doi: 10.1016/s0028-3932(01)00098-7. PMID 11640944
- [Background] Marchand Y, Friedman RB. Impaired oral reading in two atypical dyslexics: a comparison with a computational lexical-analogy model. Brain Lang. 2005 Jun;93(3):255-66. doi: 10.1016/j.bandl.2004.10.013. Epub 2004 Dec 15. PMID 15862852
- [Background] Lott SN, Sample DM, Oliver RT, Lacey EH, Friedman RB. A patient with phonologic alexia can learn to read "much" from "mud pies". Neuropsychologia. 2008 Aug;46(10):2515-23. doi: 10.1016/j.neuropsychologia.2008.04.004. Epub 2008 Apr 16. PMID 18513760
- [Background] Lott SN, Carney AS, Glezer LS, Friedman RB. Overt use of a tactile-kinesthetic strategy shifts to covert processing in rehabilitation of letter-by-letter reading. Aphasiology. 2010 Nov;24(11):1424-1442. doi: 10.1080/02687030903580333. PMID 21170161
- [Background] Lacey EH, Lott SN, Snider SF, Sperling A, Friedman RB. Multiple Oral Re-reading treatment for alexia: The parts may be greater than the whole. Neuropsychol Rehabil. 2010 Aug;20(4):601-23. doi: 10.1080/09602011003710993. Epub 2010 Jul 6. PMID 20574915
- [Background] Kurland J, Cortes CR, Wilke M, Sperling AJ, Lott SN, Tagamets MA, Vanmeter J, Friedman RB. Neural Mechanisms Underlying Learning following Semantic Mediation Treatment in a case of Phonologic Alexia. Brain Imaging Behav. 2008 Sep;2(3):147. doi: 10.1007/s11682-008-9027-2. PMID 20119495
- See also: Cognitive Neuropsychology Lab at Georgetown University Medical Center — http://explore.georgetown.edu/people/friedmar/?PageTemplateID=212